CLINICAL TRIAL: NCT04952675
Title: The Development and Clinical Application of Pneumoconiosis High Risk Early Warning Models Based on Convolutional Neural Network in Chest Radiography
Brief Title: Evaluation of Pneumoconiosis High Risk Early Warning Models
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PekingUTH-002
Record Dates: First submitted 2021-06-23; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Pneumoconiosis
Keywords: artificial intelligence; pneumoconiosis; Deep Convolutional Neural Networks; computer-aided diagnosis
MeSH Terms: conditions — Pneumoconiosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- low-risk group: Risk Index∈[0,0.5)
- high-risk group: Risk Index∈[0.5,1)

SUMMARY:
Precaution of pneumoconiosis is more important than treatment. However, the current process can't early warn the high-risk dust exposed workers until they are diagnosed with pneumoconiosis. With the feature of efficiency, impersonality and quantification, artificial intelligence is just appropriate for solving this problems. Therefore, we are aiming at adapting deep learning to develop models of pneumoconiosis intelligent detection, grade diagnosis and high risk early warning. The annotated images will be used for convolutional neural networks (CNNs) algorithm training, aiming at pneumoconiosis screening and grade diagnosis. Moreover, risk score calculated by density heat map will be used for early warning of dust-exposed workers. Then follow up of cohort will be implied to verify the validity of the risk score. By this way, the high-risk dust-exposed workers will get early intervention and better prognosis, which can obviously reduce medical burden.

DETAILED DESCRIPTION:
Pneumoconiosis, the predominant occupational disease in China and all over the world. Chest radiography is the most accessible and affordable radiological test available for the physical examination of dust-exposed workers and mass screening for pneumoconiosis. But the diagnosis process has some disadvantages, such as strong subjectivity, inefficiency, and disability of judgement of borderline lesion, etc. Besides, precaution of pneumoconiosis is more important than treatment. However, the current process can't early warn the high-risk dust exposed workers until they are diagnosed with pneumoconiosis. With the feature of efficiency, impersonality and quantification, artificial intelligence is just appropriate for solving the aforesaid problems. Up to now, there has been rare research about adapting deep learning for pneumoconiosis grade diagnosis and high risk early warning. In our previous studies, we set up a chest radiograph database, which contains more than 100,000 digital pneumoconiosis radiography images. The result of detection-system evaluation demonstrated that the accuracy in the identification of pneumoconiosis could reach 90%, with an AUC(Area Under The Curve) of 0.965 and a sensitivity of 99%. More works need to be continued. Therefore, we are aiming at adapting deep learning to develop models of pneumoconiosis intelligent detection, grade diagnosis and high risk early warning. The annotated images will be used for convolutional neural networks (CNNs) algorithm training, aiming at pneumoconiosis screening and grade diagnosis. Moreover, risk score calculated by density heat map will be used for early warning of dust-exposed workers. Then follow up of cohort will be implied to verify the validity of the risk score. By this way, the high-risk dust-exposed workers will get early intervention and better prognosis, which can obviously reduce medical burden.

ELIGIBILITY:
Inclusion Criteria:

1. workers exposed to dust;
2. have digital chest radiography

Exclusion Criteria:

1. basal pulmonary disease;
2. dimission from dust-exposed work

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: dust-exposed workers of 16 provinces of China
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
participants diagnosed as "pneumoconiosis" | before December, 31,2022
  Number of Participants diagnosed as "pneumoconiosis"
death | before December, 31,2022
  Number of Participants who dies

SECONDARY OUTCOMES:
Forced Expiratory Volume In 1s(FEV1) in % | before December, 31,2022
  Forced Expiratory Volume In 1s
arterial partial pressure of oxygen, PaO2 | before December, 31,2022
  arterial partial pressure of oxygen
modified Medical Research Council，mMRC | before December, 31,2022
  a questionnaire used to assess symptom

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Li, M.D., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided